CLINICAL TRIAL: NCT06368505
Title: A Prospective Comparative Study on the Efficacy of Ultrasound-Guided Platelet-Rich Plasma Injection Versus Hydrodissection in the Treatment of Carpal Tunnel Syndrome
Brief Title: Platelet-Rich Plasma Injection Versus Hydrodissection in the Treatment of Carpal Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osama Ahmed Elshafei (Other)
Responsible Party: Sponsor-Investigator, Osama Ahmed Elshafei, lecturer of neurology, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.24.02.2506.R1
Record Dates: First submitted 2024-04-07; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel; ultrasound guided intervention
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet rich plasma (Experimental): 3 ml PRP injection
  Interventions: Other: ultrasound guided PRP injection
- hydrodissection (Experimental): 5ml injectate
  Interventions: Other: ultrasound guided hydrodissection

INTERVENTIONS:
Other: ultrasound guided PRP injection — whole blood is initially collected in tubes that contain anticoagulants, such as citrate dextrose A to prevent platelet activation prior to its use. Then PRP is prepared by a differential centrifugation. Then 3ml of PRP will be delivered via the in-plane ulnar approach
  Arms: Platelet rich plasma
Other: ultrasound guided hydrodissection — 5ml will be injected to detach the median nerve from the TCL (2ml saline, 2ml dexamethasone and 1ml lidocaine), the injectate will be delivered via the in-plane ulnar approach, and the median nerve will be hydrodissected from its undersurface while advancing the needle among the superficial surface of the median nerve and the TCL
  Arms: hydrodissection

SUMMARY:
The goal of this clinical trial is to compare the efficacy of Ultrasound-Guided Platelet-Rich Plasma Injection versus Hydrodissection (using 2ml saline, 2ml dexamethasone and 1ml lidocaine) in the Treatment of Carpal Tunnel Syndrome. The main questions it aims to answer are:

* Which modality is more effective in reducing symptoms and improving function in patients with Carpal tunnel syndrome
* Asses safety profile of both methods

Participants will:

* Randomized to one of the two arms
* Visit the clinic 1 and 3 months after intervention
* Assessed for efficacy and safety of the intervention

DETAILED DESCRIPTION:
The medical records of patients diagnosed with carpal tunnel syndrome will be reviewed using a computerized carpal tunnel syndrome sheet including all variables for each patient assessing the symptoms and the functional condition by assessing changes in the usual daily routines. The assessment of the patients was done before and after the intervention (1 and 3 months later).

The CSA is obtained (in mm² at distal wrist crease) using ultrasound. Then the CTS grading was determined via US staging 9-13, 13-15, >15 as mild, moderate and severe respectively.

Ultrasound-Guided Intracarpal Injection. High-resolution US examination will be done by using a GE Logiq E9 with ML6-15-D Matrix linear array probe (USA). Under sterile conditions, a 25-gauge needle will be used using ulnar approach and under real time visualization the needle will be guided to the superficial ulnar aspect of the median nerve. The patients will be randomized into two groups

PRP group:

whole blood is initially collected in tubes that contain anticoagulants, such as citrate dextrose A to prevent platelet activation prior to its use. Then PRP is prepared by a differential centrifugation. Then 3ml of PRP will be delivered via the in-plane ulnar approach

Hydrodissection group:

5ml will be injected to detach the median nerve from the TCL (2ml saline, 2ml dexamethasone and 1ml lidocaine), the injectate will be delivered via the in-plane ulnar approach, and the median nerve will be hydrodissected from its undersurface while advancing the needle among the superficial surface of the median nerve and the TCL.

All patients will be observed for 30-min post-injection for possible side effects before discharge.

Outcome Measurements: All outcome assessments will be measured at 1 and 3 months after intervention.

Primary Outcome Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) and The visual analog scale (VAS) to assess the efficacy of interventions Secondary Outcome The cross-sectional area (CSA) of the Median nerve will be measured by the same US machine, Measurements were repeated 3 times and averaged for further

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed clinically as carpal tunnel syndrome with at least 3 months of symptoms and confirmed electro-physiologically as carpal tunnel syndrome

Exclusion Criteria:

* Onset of carpal tunnel syndrome during pregnancy
* Co-existence of brachial plexopathy or thoracic outlet syndrome by clinical examination
* Previous carpal tunnel decompressive surgery or corticosteroid injection in carpal tunnel
* Patients with infection or local edema at the site of injection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-06-16 (Estimated); Study Completion 2024-07-16 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) | before the intervention,1 and 3 months after intervention
  Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) is a patient-based questionnaire, consists of two main scales:
  Symptom Severity Scale (SSS): Measures the severity of symptoms related to CTS. Functional Status Scale (FSS): Assesses functional limitations caused by CTS. Each scale contains several items, and patients rate their symptoms or functional difficulties on a scale from 1 to 5.
  A score of 1 indicates no symptoms or functional difficulty. A score of 5 represents maximum symptoms or inability to perform the task1.
  Interpretation:
  Higher scores on both scales indicate worse symptoms or greater functional impairment due to CTS.
The visual analog scale (VAS) | before the intervention,1 and 3 months after intervention
  The Visual Analogue Scale (VAS) is a simple assessment tool used to measure pain intensity.
  The VAS consists of a straight horizontal line, usually 10 centimetres (cm) in length.
  One end of the line represents "no pain," while the other end represents "the worst pain ever experienced." Patients are asked to rate their current level of pain by placing a mark on the line.
  Using a ruler, the score is determined by measuring the distance (in millimetres) from the "no pain" anchor to the patient's mark.
  The resulting score ranges from 0 to 100, with a higher score indicating greater pain intensity.

SECONDARY OUTCOMES:
The cross-sectional area (CSA) of the Median nerve | before the intervention and 3 months after intervention
  Using the ultrasound, the CSA is obtained (in mm² at distal wrist crease) by utilizing the tracing function on the US machine by direct tracing around the inner margin of the epineurium but with no weaving in between each fascicle. Measurements were repeated three times and average value was used for statistical evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR